CLINICAL TRIAL: NCT04300647
Title: A Phase II, Safety, and Efficacy Study of Tiragolumab Plus Atezolizumab and Atezolizumab Monotherapy in Patients With Metastatic and/or Recurrent PD-L1-Positive Cervical Cancer
Brief Title: A Study of Tiragolumab Plus Atezolizumab and Atezolizumab Monotherapy in Participants With Metastatic and/or Recurrent PD-L1-Positive Cervical Cancer
Acronym: SKYSCRAPER-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO42017; 2019-004895-21 (EudraCT Number)
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Tiragolumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tiragolumab plus Atezolizumab (Experimental): Participants will receive tiragolumab and atezolizumab until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab
- Atezolizumab (Experimental): Participants will receive atezolizumab monotherapy until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Tiragolumab — Tiragolumab at a fixed dose of 600 milligrams (mg) will be administered by intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Other Names: RO7092284
  Arms: Tiragolumab plus Atezolizumab
Drug: Atezolizumab — Atezolizumab at a fixed dose of 1200 mg will be administered by IV infusion Q3W on Day 1 of each 21-day cycle.
  Other Names: RO5541267; Tecentriq

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tiragolumab in combination with atezolizumab and atezolizumab monotherapy in patients with programmed death-ligand 1 (PD-L1)-positive cervical cancer (metastatic and/or recurrent).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or persistent squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix after progression on or after 1-2 lines of prior systemic chemotherapy in the metastatic/recurrent setting that is not amenable to curative treatment with systemic chemotherapy, surgery, and/or radiotherapy
* Radiologically-measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance Status of 0 or 1
* Cervical cancer tissue for study analysis (archival or fresh biopsy specimen)
* Life expectancy of at least 12 weeks
* Adequate hematologic and organ function
* Female of childbearing potential must be willing to comply with adequate contraception

Exclusion Criteria:

* Treatment with investigational therapy with therapeutic intent within 28 days prior to randomization
* Active or untreated central nervous system (CNS) or brain metastases
* Active or history of autoimmune disease or immune deficiency
* Active tuberculosis
* Known, clinically significant liver disease
* Severe infection per investigator judgement at the time of randomization or any active infection that, in the opinion of the investigator, could impact patient safety
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-CTLA-4, anti-TIGIT, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to randomization
* Treatment with systemic immunosuppressive medications within 1 week prior to randomization or anticipation of need for systemic immunosuppressive medication during study
* Pregnant or breastfeeding woman
* Known hypersensitivity to any component of the tiragolumab or atezolizumab formulations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (56):
- United States (4):
  - Arizona Oncology Associates, Phoenix, Arizona
  - Kaiser Permanente - Irvine, Irvine, California
  - Augusta University, Augusta, Georgia
  - Oncology Associates of Oregon, P.C, Eugene, Oregon
- Mater Misericordiae Limited, South Brisbane, Queensland, Australia
- Brazil (5):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital de Caridade de Ijui, Ijuí, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
- Canada (5):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- Costa Rica (2):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
- France (5):
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Régional de Lutte Contre Le Cancer Val D'aurelle Paul Lamarque, Montpellier
  - ICO - Site René Gauducheau, Saint-Herblain
  - Gustave Roussy, Villejuif
- Italy (3):
  - Istituto Tumori Napoli, Napoli, Campania
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Istituto Europeo Di Oncologia, Milan, Lombardy
- Christus Muguerza Clinica Vidriera, Monterrey, Nuevo León, Mexico
- Panama (2):
  - Centro Oncológico de Panamá, Panama City
  - The Panama Clinic, Panama City
- Clinica Ricardo Palma, San Isidro, Peru
- Poland (4):
  - Szpital Morski im.PCK, Gdynia
  - Narodowy Inst.Onkol.im.Sklodowskiej-Curie Panstw.Inst.Bad Gliwice, Gliwice
  - Wielkopolskie Centrum Onkologii im. M. Sklodowskiej-Curie, Poznan
  - Narodowy Instytut Onkologii im. M.Sklodowskiej-Curie, Warsaw
- Russia (5):
  - MEDSI Clinical Hospital on Pyatnitsky Highway, Moscow, Moscow Oblast
  - Chelyabisnk regional clinical center for oncology and nuclear medicine, Chelyabinsk, Sverdlovsk Oblast
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan', Tatarstan Republic
  - Tomsk scientific research institute of oncology SO RAMN, PAD, Tomsk
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
- South Korea (7):
  - Keimyung University Dongsan Hospital, Daegu
  - Korea Cancer Center Hospital of Korea Institute of Radiological and Medical Sciences, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Medical Foundation, Linkou Branch, Taoyuan
- Maharaj Nakorn Chiang Mai Hospital, Muang, Thailand
- United Kingdom (2):
  - University College London Hospital, London
  - Sarah Cannon Research Institute, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Salani R, McCormack M, Kim YM, Ghamande S, Hall SL, Lorusso D, Barraclough L, Gilbert L, Guzman Ramirez A, Lu CH, Sabatier R, Colombo N, Hu Y, Krishnan V, Molinero L, Feng Y, Kim N, Castro M, Lin YG, Monk BJ. A non-comparative, randomized, phase II trial of atezolizumab or atezolizumab plus tiragolumab for programmed death-ligand 1-positive recurrent cervical cancer (SKYSCRAPER-04). Int J Gynecol Cancer. 2024 Aug 5;34(8):1140-1148. doi: 10.1136/ijgc-2024-005588. PMID 38858106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 59 centers in 17 countries. The study enrolled 172 participants of whom 171 were included in the Treated Population reported here. The study is ongoing. Data up to primary completion date is reported here.
Pre-assignment Details: Subjects with PDL1-positive cervical cancer were randomized in a 3:1 ratio to receive either atezolizumab plus tiragolumab or atezolizumab monotherapy with the use of a stratified permuted-block randomization based on Eastern Cooperative Oncology Group (ECOG) Performance Status, prior use of chemoradiotherapy or radiotherapy, and treatment history.
Groups:
- Atezolizumab: Participants received atezolizumab monotherapy until disease progression, loss of clinical benefit, or unacceptable toxicity as determined by the investigator.
- Tiragolumab Plus Atezolizumab: Participants received tiragolumab and atezolizumab until disease progression, loss of clinical benefit, or unacceptable toxicity as determined by the investigator.
- Post Crossover Tiragolumab Plus Atezolizumab: After unequivocal progressive disease had been recorded during atezolizumab monotherapy, crossover was allowed from the atezolizumab monotherapy arm to the tiragolumab plus atezolizumab arm at the discretion of the investigator and after consultation with the Medical Monitor.
Period: Pre-Crossover
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab | Post Crossover Tiragolumab Plus Atezolizumab
Started (Treated Population) | 45 | 126 | 0
Completed | 0 | 0 | 0
Not Completed | 45 | 126 | 0
Not completed — Death | 19 | 58 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0
Not completed — On-going in Study | 24 | 61 | 0
Period: Post-Crossover
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab | Post Crossover Tiragolumab Plus Atezolizumab
Started | 0 | 0 | 13
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 13
Not completed — Death | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — On-going in Study | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab | Total
Number analyzed (Participants) | 45 | 126 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (11.8) | 50.8 (11.8) | 50.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 126 | 171
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 18 | 25
  Not Hispanic or Latino | 32 | 81 | 113
  Unknown or Not Reported | 6 | 27 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 6 | 16 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 28 | 79 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 27 | 34
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status grades 0 or 1 were used for stratified randomization. Grade 0: Fully active, able to carry on all pre-disease performance without restriction. Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light house work, office work).
  Participants
    ECOG Performance Status 0 | 23 | 55 | 78
    ECOG Performance Status 1 | 22 | 71 | 93
Prior Use of Chemoradiotherapy or Radiotherapy [Count of Participants; unit: Participants] — Prior use of chemotherapy or radiotherapy "yes" or "no" was used for stratified randomization.
  Participants
    Yes | 36 | 98 | 134
    No | 9 | 28 | 37
Treatment History [Count of Participants; unit: Participants] — Treatment history of recurrent versus persistent disease was used for stratified randomization.
  Participants
    Recurrent Disease | 26 | 65 | 91
    Persistent Disease | 19 | 61 | 80

OUTCOME MEASURES:

1. Primary Outcome: Independent Review Committee (IRC)-Assessed Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a complete response (CR) or a partial response (PR) on two consecutive occasions >/=4 weeks apart, as determined by the IRC according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. The study enrolled patients with measurable disease as determined by the investigator. Participants found to have non-measurable disease at baseline according to RECIST v1.1 (through IRC assessment or Protocol Deviations) were only considered responders if they achieved a CR.
Time Frame: From randomization up to approximately 17 months
Population: The Treated Population was defined as all randomized participants that received at least any dose of study treatment. Participants are grouped according to the actual treatment received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab
Number analyzed (Participants) | 45 | 126
percentage of participants | 15.6 [6.5 to 29.5] | 19.0 [12.6 to 27.0]

2. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 36 months
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: IRC-Assessed Duration of Response (DOR)
Description: DOR is defined for participants who had an objective response as the time from the first occurrence of a documented objective response (CR or PR) to the date of progressive disease (PD) or death from any cause (whichever occurred first), as determined by the IRC according to RECIST v1.1. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline). The study enrolled patients with measurable disease as determined by the investigator. Participants found to have non-measurable disease at baseline according to RECIST v1.1 (through IRC assessment or Protocol Deviations) were only considered responders if they achieved a CR.
Time Frame: First occurrence of a documented objective response to the date of disease progression or death from any cause, whichever occurs first (up to approximately 17 months)
Population: The Treated Population was defined as all randomized participants that received at least any dose of study treatment. Participants are grouped according to the actual treatment received. DOR was assessed in participants with an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab
Number analyzed (Participants) | 7 | 24
months | NA [6.5 to NA] — NA: the median duration of ORR was not reached due to low number of participants with events. | 11.8 [6.7 to NA] — Na: not estimable due to low number of participants with events.

4. Secondary Outcome: IRC-Assessed Disease Control Rate (DCR)
Description: Disease control rate is defined as the percentage of participants with a CR, PR, or stable disease (SD), as determined by the IRC according to RECIST v1.1. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. SD: neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. Participants were classified as SD only if SD was observed on two consecutive assessments >/= 6 weeks apart. The study enrolled patients with measurable disease as determined by the investigator. Participants found to have non-measurable disease at baseline according to RECIST v1.1 (through IRC assessment or Protocol Deviations) were only considered responders if they achieved a CR.
Time Frame: From randomization up to approximately 17 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab
Number analyzed (Participants) | 45 | 126
percentage of participants | 20.0 [9.6 to 34.6] | 31.0 [23.0 to 39.8]

5. Secondary Outcome: Investigator-Assessed Best Clinical Response (BCR) Rate
Description: BCR is defined as the percentage of participants with a CR, PR, or SD, as determined by the investigator. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. SD: neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. Participants were classified as SD only if SD was observed on two consecutive assessments >/= 6 weeks apart.
Time Frame: From randomization up to approximately 17 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab
Number analyzed (Participants) | 45 | 126
percentage of participants | 33.3 [20.0 to 49.0] | 44.4 [35.6 to 53.6]

6. Secondary Outcome: Investigator-Assessed Duration of BCR
Description: Duration of BCR is defined for BCR responders as the time from the first occurrence of a documented response (CR, PR, or SD) to the date of PD or death from any cause (whichever occurred first), as clinically determined by the investigator according to RECIST v1.1. CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. SD: neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. Participants were classified as SD only if SD was observed on two consecutive assessments >/= 6 weeks apart. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline).
Time Frame: First occurrence of a documented clinical response to the date of disease progression or death from any cause, whichever occurs first (up to approximately 17 months)
Population: The Treated Population was defined as all randomized participants that received at least any dose of study treatment. Participants are grouped according to the actual treatment received. Duration of BCR was assessed in participants with a clinical response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab
Number analyzed (Participants) | 15 | 56
months | 7.0 [5.6 to NA] — NA: not estimable due to low number of events. | 5.5 [4.2 to 8.7]

7. Secondary Outcome: IRC-Assessed Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first occurrence of PD or death from any cause (whichever occurred first), as determined by the IRC according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline).
Time Frame: From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 17 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab
Number analyzed (Participants) | 45 | 126
months | 1.9 [1.5 to 3.0] | 2.8 [1.7 to 4.1]

8. Secondary Outcome: IRC-Assessed PFS Rate at 6 Months
Description: PFS rate is defined as the percentage of participants that were event free, as determined by the IRC according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline).
Time Frame: 6 months
Population: The Treated Population was defined as all randomized participants that received at least any dose of study treatment. Participants are grouped according to the actual treatment received. Overall number analyzed are number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specified timepoints
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab
Number analyzed (Participants) | 9 | 34
percentage of participants | 21.50 [9.06 to 33.94] | 30.56 [22.29 to 38.83]

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time of randomization to death from any cause.
Time Frame: From randomization to death from any cause (up to approximately 17 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab
Number analyzed (Participants) | 45 | 126
months | 10.6 [7.4 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events. | 11.0 [9.6 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.

10. Secondary Outcome: OS Rate at 6 Months and 12 Months
Description: Reported here are the percentages of participants who were still alive at 6 months and 12 months.
Time Frame: 6 months, 12 months
Population: The Treated Population was defined as all randomized participants that received at least any dose of study treatment. Overall number analyzed are number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specified timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab
Number analyzed (Participants) | 26 | 86
percentage of participants
  6 Months | 69.49 [55.52 to 83.47] | 73.56 [65.69 to 81.44]
  12 Months: number analyzed (Participants) | 5 | 16
  12 Months | 37.88 [17.38 to 58.38] | 47.19 [36.63 to 57.76]

11. Other Pre Specified Outcome: Minimum Serum Concentration (Cmin) of Tiragolumab
Time Frame: Pre dose: Day 1 of Cycles 2, 3, 4, 8, 12 and 16
Reporting Status: Not Posted, anticipated posting 2025-12

12. Other Pre Specified Outcome: Maximum Serum Concentration (Cmax) of Tiragolumab
Time Frame: Cycle 1 Day 1 at 30 minutes post-dose
Reporting Status: Not Posted, anticipated posting 2025-12

13. Other Pre Specified Outcome: Cmin of Atezolizumab
Time Frame: Pre dose: Day 1 of Cycles 2, 3, 4, 8, 12 and 16
Reporting Status: Not Posted, anticipated posting 2025-12

14. Other Pre Specified Outcome: Cmax of Atezolizumab
Time Frame: Day 1 of Cycle 1 at 30 minutes post-dose
Reporting Status: Not Posted, anticipated posting 2025-12

15. Other Pre Specified Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Tiragolumab
Description: Participants were classified as treatment-emergent ADA-positive if they were ADA negative at baseline or missing data but developed an ADA response following study drug administration (treatment-induced ADA response) or if they were ADA-positive at baseline and the titre of one or more post-baseline samples was at least 4-fold greater (i.e., ≥ 0.60 titre units) than the titre of the baseline sample (treatment-enhanced ADA response).
Time Frame: Predose on Day 1 of Cycles (each cycle is 21 days) 1, 2, 3, 4, 8, 12 and 16
Reporting Status: Not Posted, anticipated posting 2025-12

16. Other Pre Specified Outcome: Percentage of Participants With ADAs to Atezolizumab
Description: as for outcome 15
Time Frame: Predose on Day 1 of Cycles (each cycle is 21 days) 1, 2, 3, 4, 8, 12 and 16
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: From initiation of study treatment up to 90 days after last dose (approximately 17 months) Data collection is ongoing, the Adverse Events section will be updated one year after study completion date.
Description: Treated Population=all randomized participants that received at least one dose of study treatment. Participants are grouped according to the actual treatment received. Participants crossing over from atezolizumab to tiragolumab plus atezolizumab arm are represented separately post crossover. All AEs: reported until 30 days after the last study dose/start of new systemic anti-cancer therapy. SAEs & AEs of special interest: reported up to 90 days after last study dose.
Arm/Group | Atezolizumab | Tiragolumab Plus Atezolizumab | Post Crossover Tiragolumab Plus Atezolizumab
All-Cause Mortality (participants affected / at risk) | 19/45 | 58/126 | 3/13
Serious Adverse Events (participants affected / at risk) | 12/45 | 37/126 | 0/13
Other Adverse Events (participants affected / at risk) | 36/45 | 108/126 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=45) | Tiragolumab Plus Atezolizumab (N=126) | Post Crossover Tiragolumab Plus Atezolizumab (N=13)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (6) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (4) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 4 (4) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab (N=45) | Tiragolumab Plus Atezolizumab (N=126) | Post Crossover Tiragolumab Plus Atezolizumab (N=13)
Anaemia (Blood and lymphatic system disorders) | 9 (20) | 39 (86) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (4) | 5 (14) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 2 (4) | 7 (14) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (6) | 7 (14) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 17 (40) | 3 (6)
Abdominal pain upper (Gastrointestinal disorders) | 3 (6) | 4 (8) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (10) | 13 (36) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (6) | 17 (48) | 2 (4)
Nausea (Gastrointestinal disorders) | 5 (10) | 25 (60) | 2 (4)
Vomiting (Gastrointestinal disorders) | 7 (14) | 18 (46) | 1 (2)
Asthenia (General disorders) | 6 (12) | 22 (52) | 1 (2)
Chills (General disorders) | 2 (4) | 4 (10) | 1 (2)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 3 (6) | 22 (58) | 1 (2)
Oedema peripheral (General disorders) | 3 (8) | 10 (22) | 1 (2)
Pyrexia (General disorders) | 6 (18) | 20 (46) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (2)
Urinary tract infection (Infections and infestations) | 2 (4) | 16 (48) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (10) | 10 (22) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (8) | 8 (16) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 9 (20) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 8 (16) | 2 (4)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 3 (6) | 5 (12) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 2 (4) | 2 (4)
Blood magnesium increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood sodium decreased (Investigations) | 0 (0) | 1 (2) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 1 (2) | 1 (2)
Weight decreased (Investigations) | 1 (2) | 9 (18) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (6) | 18 (38) | 1 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 10 (22) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (14) | 15 (42) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 10 (24) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6) | 5 (10) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 6 (14) | 1 (2)
Headache (Nervous system disorders) | 2 (4) | 12 (32) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 8 (16) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (4) | 7 (14) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (2) | 7 (16) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 8 (16) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (10) | 5 (12) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 23 (60) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 11 (22) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT04300647/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT04300647/SAP_001.pdf